CLINICAL TRIAL: NCT04780230
Title: Modulation of Primary Motor Cortex to Enhance Treatment of Dysarthria Post-stroke
Brief Title: Non-invasive Brain Stimulation to Enhance Treatment of Dysarthria Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The University of Hong Kong (Other); Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Min Wong, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRESC201906
Record Dates: First submitted 2021-02-19; First posted 2021-03-03 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Dysarthria; Stroke
MeSH Terms: conditions — Dysarthria; Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real tDCS (Experimental): A total of 60 Cantonese-speaking post-stroke patients who are suffering from dysarthria will be recruited and randomly divided into real tDCS and sham groups.
  Interventions: Device: tDCS active
- sham tDCS (Sham Comparator): A total of 60 Cantonese-speaking post-stroke patients who are suffering from dysarthria will be recruited and randomly divided into real tDCS and sham groups.
  Interventions: Device: tDCS sham

INTERVENTIONS:
Device: tDCS active — An anodal high-definition tDCS of 2 mA lasting for 20 minutes will be delivered to the orofacial area of the primary motor cortex (SM1) during speech therapy.
  Arms: real tDCS
Device: tDCS sham — An anodal high-definition tDCS of 2 mA lasting for 30 seconds will be delivered to the orofacial area of the primary motor cortex (SM1) during speech therapy.
  Arms: sham tDCS

SUMMARY:
The proposed study aims to determine if transcranial direct current stimulation can enhance the effect of speech therapy in post-stroke patients with dysarthria.

DETAILED DESCRIPTION:
A total of 60 Cantonese-speaking post-stroke patients who are suffering from dysarthria will be recruited and randomly divided into real tDCS and sham groups. All the participants will receive individualized speech therapy based on the results of their speech assessment.

For the real tDCS group, an anodal high-definition tDCS of 2 milliamperes (mA) lasting for 20 minutes will be delivered to the orofacial area of the primary motor cortex (SM1) during speech therapy. For the sham tDCS group, stimulation given during speech therapy will only last for 30 seconds in order to cause a similar sensation on the scalp as the real stimulation group. There will be a total of 10 daily sessions during a 2-week period.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese-speaking adults who had their first stroke and have suffered dysarthria post-stroke.
* Both acute and chronic stroke participants will be recruited.

Exclusion Criteria:

* Individuals with a personal or family history of epilepsy or seizures;
* Individuals with a history of another neurological condition (which is not a result from the initial stroke);
* Individuals with a history of speech disorders, voice disorders, oro-maxillo-facial surgery involving the tongue and/or lip, severe cognitive impairment, severe aphasia;
* In an unstable or serious medical condition;
* Have a cardiac implant metallic foreign body implant and/or any medications that lower neural thresholds (e.g. antidepressants, neuroleptic agents, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Perceptual speech assessments | Change Before and After tDCS Stimulation at immediately post-treatment, 1-month and 3-month post treatment
  All participants will be required to produce a sustained vowel /a/, repeat some syllables (i.e., /pa/, /ta/, /ka/ and /pataka/), read a standard Chinese paragraph and have a 1-2 mins conversation with the researcher.
Communication effectiveness measures | Change Before and After tDCS Stimulation at immediately post-treatment, 1-month and 3-month post treatment
  The Modified Communication Effectiveness Index (CETI-M) is a 10-item patient-reported measure of change in functional communication ability.

SECONDARY OUTCOMES:
Kinematic Measurements | Change Before and After tDCS Stimulation at immediately post-treatment, 1-month and 3-month post treatment
  The lip and tongue function during speech production will be traced real time and objectively using the 3D-Electromagnetic Articulography (EMA, AG501-system).
Acoustic measurements | Change Before and After tDCS Stimulation at immediately post-treatment, 1-month and 3-month post treatment
  Acoustic measurements will be obtained from both sustained vowel phonation and connected speech.
Quality of Life measurement | Change Before and After tDCS Stimulation at immediately post-treatment, 1-month and 3-month post treatment
  The Chinese version of The Quality of Life of the Dysarthric Speaker (QOL-DyS) questionnaire will be used to assess participants' subjective speech related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Min Ney Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No